CLINICAL TRIAL: NCT06812416
Title: Effectiveness of Qualia NAD+ Supplementation on Intracellular NAD Levels: a Randomized Double-Blind Parallel Trial
Brief Title: Effectiveness of Qualia NAD+ Supplementation on NAD Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NHC-003
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Intracellular NAD+ Levels
Keywords: NAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qualia NAD+ (Active Comparator): Qualia NAD+
  Interventions: Dietary Supplement: Qualia NAD+
- Placebo (Placebo Comparator): Rice Flour Placebo
  Interventions: Dietary Supplement: Rice Flour Placebo

INTERVENTIONS:
Dietary Supplement: Qualia NAD+ — Qualia NAD+
  Arms: Qualia NAD+
Dietary Supplement: Rice Flour Placebo — Rice Flour Placebo
  Arms: Placebo

SUMMARY:
The current study is designed as a randomized double-blind placebo-controlled parallel trial. It aims to investigate the efficacy of Qualia NAD+ on intracellular NAD levels in blood samples (primary outcomes) and health-related quality of life (secondary outcomes) in an adult population experiencing moderate to severe joint pain between ages of 40 and 65 years.

ELIGIBILITY:
Inclusion criteria:

Provide voluntary, written, informed consent to participate in the study Agree to provide a valid cell phone number and are willing to receive communications through text.

Healthy male and female participants between the ages of 40-65 years of age. Willingness to complete questionnaires, records, and diaries associated with the study.

Willing to not consume any supplements, energy drinks/shots, or other products containing any form of supplemental vitamin B3 (e.g., niacin, niacinamide, nicotinamide ribosome, NMN) starting about 2 weeks prior to the baseline NAD fingerstick test and continuing through the intervention period.

Willing to not begin taking any new supplements during the study period, and to continue taking any supplements they are currently using regularly (with the exception of vitamin B3 containing supplements).

Willing to self-administer the intracellular NAD fingerstick test kit at home for both a baseline and post-intervention blood sample, and to complete a release form that gives NHC access to the results of these tests.

Exclusion criteria:

Women who are pregnant, breastfeeding, or planning to become pregnant during the trial Known food intolerances/allergy to any ingredients in the product Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer Having had a significant cardiovascular event in the past 6 months Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines On immunosuppressive therapy Individuals who were deemed incompatible with the test protocol Adults lacking capacity to consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Intracellular NAD+ Levels | Baseline and day 28

SECONDARY OUTCOMES:
Aging Male/Female Symptom scale | Baseline, day 14, and day 28
RAND SF-36 | Baseline, day 14, and day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Remote Study, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No